CLINICAL TRIAL: NCT00232310
Title: Double Blind Placebo Controlled Dose Ranging Study of the Efficacy and Safety of SSR149744C 300 or 600 mg for the Conversion of Atrial Fibrillation / Flutter
Acronym: CORYFEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI5760
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Electric Countershock
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — celivarone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: CELIVARONE (SSR149744C)

SUMMARY:
Double blind study to assess versus placebo the efficacy of SSR149744C for the conversion of atrial fibrillation/flutter to sinus rhythm at the time of the planned electrical cardioversion.

DETAILED DESCRIPTION:
This is a dose ranging multicenter, multinational, randomized, double blind, placebo controlled, parallel arm study. Patients with AF/AFL will be randomized to one of two doses of SSR149744C.

The efficacy of SSR149744C will be based on the proportion of patients converting to normal sinus rhythm at the end of the treatment period (48 hours post first dose).

Patients will receive the study drug on D1 and D2. Patients not converting pharmacologically to sinus rhythm will undergo an electrical cardioversion on D3.

ELIGIBILITY:
Inclusion Criteria:

* AF/AFL for >72 hours and documented by 2 12-lead ECGs separated by at least 72 hours and indication for electrical cardioversion of the current AF/AFL episode as judged by the investigator.

Exclusion Criteria:

MAIN CRITERIA (non-exhaustive list):

* Women of childbearing potential without adequate birthcontrol, Pregnant Women, Breastfeeding women, conditions which increase the risk of severe antiarrhythmic drug side effects, permanent pacemaker, permanent AF/AFL, contraindication to anticoagulant, severe left ventricular dysfunction, severe associated conditions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-10; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the rate of conversion to sinus rhythm documented by ECG just before the planned electrical cardioversion on D3 i.e. after 48 hours following the first study drug administration.

SECONDARY OUTCOMES:
The secondary efficacy endpoint will be the mean ventricular rate during AF/AFL on the 12-lead ECG performed just before the planned electrical cardioversion on D3 i.e. after 48 hours following the first study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (9):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal

REFERENCES:
- [Result] Khitri AR, Aliot EM, Capucci A, Connolly SJ, Crijns H, Hohnloser SH, Kulakowski P, Roy D, Radzik D, Kowey PR. Celivarone for maintenance of sinus rhythm and conversion of atrial fibrillation/flutter. J Cardiovasc Electrophysiol. 2012 May;23(5):462-72. doi: 10.1111/j.1540-8167.2011.02234.x. Epub 2011 Dec 15. PMID 22171925